CLINICAL TRIAL: NCT03516890
Title: Management of Spontaneous Ruptured Hepatocellular Carcinoma - Partial Hepatectomy and Prognosis: A Retrospective Study
Brief Title: Management of Spontaneous Ruptured Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Professor, Huazhong University of Science and Technology
Other Study IDs: Chenxp010
Record Dates: First submitted 2018-04-04; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Rupture, Spontaneous; Rupture Liver; Hepatocellular Carcinoma
Keywords: Partial hepatectomy; Emergency; Staged; Peritoneal dissemination; Propensity score matching
MeSH Terms: conditions — Rupture, Spontaneous; Carcinoma, Hepatocellular; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Partial hepatectomy — Partial hepatectomy was comprised of single or multiple liver resections aiming to excise all macroscopic tumors.

SUMMARY:
To investigate the best treatment for hepatocellular carcinoma rupture

DETAILED DESCRIPTION:
To investigate the best treatment for hepatocellular carcinoma rupture, transcatheter arterial embolization or partial hepatectomy. Furthermore, to discuss the choice of emergency or staged hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed as hepatocellular carcinoma with tumor rupture; with complete data and without loss of follow-up

Exclusion Criteria:

* Without complete data; with loss of follow-up; not hepatocellular carcinoma based on pathological diagnosis

Ages: 15 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From January 2005 to June 2015, all patients complied with the criteria mentioned above who received partial hepatectomy or non-surgical at our center were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Overall survival of all patients | 5 years
  Overall survival difference between the partial hepatectomy group and the non-surgical group

SECONDARY OUTCOMES:
Postoperative peritoneal dissemination | 5 years
  Postoperative peritoneal dissemination diagnosed by imaging examination
Recurrence-free survival of all patients | 5 years
  Recurrence-free survival difference between the partial hepatectomy group and the non-surgical group
Overall survival of partial hepatectomy patients | 5 years
  Overall survival difference between the emergency partial hepatectomy group and the staged partial hepatectomy group
Recurrence-free survival of partial hepatectomy patients | 5 years
  Recurrence-free survival difference between the emergency partial hepatectomy group and the staged partial hepatectomy group
Overall survival of staged partial hepatectomy patients | 5 years
  Overall survival difference between the staged early partial hepatectomy group and the staged late partial hepatectomy group
Recurrence-free of staged partial hepatectomy patients | 5 years
  Recurrence-free survival difference between the staged early partial hepatectomy group and the staged late partial hepatectomy group

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-ping Chen, PHD, Study Chair — Huazhong University of Science and Technology

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT03516890/SAP_000.pdf